CLINICAL TRIAL: NCT04258527
Title: A Phase 1, Open-Label, Pharmacokinetic(PK), Pharmacodynamics(PD) and Safety Study of Pemigatinib in Patients With Advanced Malignancies With FGF/FGFR Alterations
Brief Title: Phase 1 Study of Pemigatinib in Patients With Advanced Malignancies With FGF/FGFR Alterations
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIBI375A101
Record Dates: First submitted 2020-01-20; First posted 2020-02-06 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Solid Tumor
MeSH Terms: interventions — pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with advanced malignancies with FGF/FGFR alterations (Experimental)
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Pemigatinib — Pemigatinib will be self-administered as at 13.5mg a QD oral treatment on a 2-week-on therapy and 1-week-off therapy schedule.

SUMMARY:
This is a phase 1 study to investigate the characteristics of PK, PD and safety in subjects with advanced malignancies with FGF/FGFR alterations.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 18 or older.
2. Histologically or cytologically confirmed malignancy which was considered to be surgically unresectable advanced, relapse or metastatic .
3. Radiographically measurable disease per RECIST v 1.1
4. Documentation of FGF/FGFR alteration..
5. Documented disease progression after standard therapy ,or no standard therapy available.
6. ECOG performance status of 0~1.
7. Life expectancy ≥12 weeks

Exclusion Criteria:

1. Prior receipt of a selective FGFR inhibitor.
2. History of calcium and phosphate hemostasis disorder or systemic mineral imbalance with ectopic calcification of softy tissues ( exception: skin, kidney, tendons or vessels due to injury, disease, and aging, in the absence of systemic mineral imbalance).
3. Currently evidence of clinically significant corneal or retinal disorder confirmed by ophthalmologic examination.
4. Use of any potent CYP3A4 inhibitors or inducers within 14 days or 5 half-lives, whichever is shorter, before the first dose of study drug. Topical ketoconazole will be allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-03-26 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) during the dosing interval and Cmin of Pemigatinib as monotherapy | Day 1 to Day 16
Time to maximum plasma concentration (Tmax) of Pemigatinib as monotherapy | Day 1 to Day 16
Area under the single-dose plasma concentration-time curve (AUC0-t) of Pemigatinib as monotherapy | Day 1 to Day 16

SECONDARY OUTCOMES:
Safety of pemigatinib as monotherapy as assessed by the frequency, duration, and severity of adverse events | From screening through 30-35 days after end of treatment, up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of Tianjin Medical University, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deng T, Zhang L, Shi Y, Bai G, Pan Y, Shen A, Han X, Yang Z, Chen M, Zhou H, Luo Y, Zheng S, Ba Y. Pharmacokinetics, pharmacodynamics and efficacy of pemigatinib (a selective inhibitor of fibroblast growth factor receptor 1-3) monotherapy in Chinese patients with advanced solid tumors: a phase i clinical trial. Invest New Drugs. 2023 Dec;41(6):808-815. doi: 10.1007/s10637-023-01396-x. Epub 2023 Oct 27. PMID 37889382